CLINICAL TRIAL: NCT03829852
Title: Investigate the Real-life Treatment Outcome of Regorafenib in Treating mCRC Patients
Brief Title: Regorafenib in Taiwan Metastatic Colorectal Cancer (mCRC) Patients
Status: Completed | Type: Observational
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Collaborators: Chang Gung Memorial Hospital (Other); Koo Foundation Sun Yat-Sen Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-12-013BC
Record Dates: First submitted 2019-01-19; First posted 2019-02-04 (Actual); Last update posted 2021-07-23 (Actual); Status verified 2021-07

CONDITIONS: Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — regorafenib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Regorafenib — Treatment was performed based on physician's discretion

SUMMARY:
Regorafenib is currently the standard of care for refractory mCRC patients. Pivotal studies of regorafenib have proven the efficacy and safety, with a 28-day cycle (21 days on, 7 days off) and 160 mg dose given once daily.

In the clinic, patients often have some complicated condition. This study aims to perform retrospective medical chart review of mCRC patients who received regorafenib treatment in two medical centers in Taiwan to examine treatment effectiveness in the routine clinical practice setting.

ELIGIBILITY:
Inclusion Criteria:

* mCRC patients who received at least one dose of regorafenib treatment

Exclusion Criteria:

* <=20 y/o
* Patients who did not receive regorafenib treatment will be excluded from the analysis
* Patients with incomplete medical records that are deemed ineligible for analysis by investigator

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: mCRC patients who received regorafenib treatment in Taipei Veterans General Hospital and Chang Gung Memorial Hospital Linkou, Taiwan
Sampling Method: Non-Probability Sample
Enrollment: 716 (Actual)
Dates: Start 2019-02-11 (Actual); Primary Completion 2020-12-08 (Actual); Study Completion 2020-12-08 (Actual)

PRIMARY OUTCOMES:
Effectiveness of regorafenib use in routine clinical practice setting, assessed by overall survival (OS) | through study completion, estimated 2 years
  months
Effectiveness of regorafenib use in routine clinical practice setting, assessed by progression free survival (PFS) | through study completion, estimated 2 years
  months
Effectiveness of regorafenib use in routine clinical practice setting, assessed by time to progression (TTP) | through study completion, estimated 2 years
  months
Effectiveness of regorafenib use in routine clinical practice setting, assessed by tumor response | through study completion, estimated 2 years
  percentage

SECONDARY OUTCOMES:
Safety of regorafenib use in routine clinical practice setting, assessed by incidence of adverse events (AEs) | through study completion, estimated 2 years
  percentage
Safety of regorafenib use in routine clinical practice setting, assessed by initial dose | through study completion, estimated 2 years
  percentage
Safety of regorafenib use in routine clinical practice setting, assessed by dose intensity during the first 2 cycles | through study completion, estimated 2 years
  percentage
Eligibility of subsequent therapies and the outcome, assessed by type of treatment (anti-epithelial growth factor receptor [EGFR], anti-vascular endothelial growth factor [VEGF], and/or chemotherapy agents) | through study completion, estimated 2 years
  percentage
Eligibility of subsequent therapies and the outcome, assessed by treatment duration | through study completion, estimated 2 years
  months
Eligibility of subsequent therapies and the outcome, assessed by PFS | through study completion, estimated 2 years
  months

OTHER OUTCOMES:
Exploratory outcome:Clinical markers/ biomarkers as the potential predictive factor for regorafenib treatment outcome in overall cohort and long-term responders, assessed by patient characteristics | through study completion, estimated 2 years
  correlation
Exploratory outcome:Clinical markers/ biomarkers as the potential predictive factor for regorafenib treatment outcome in overall cohort and long-term responders, assessed by changes in carcinoembryonic antigen (CEA) levels | through study completion, estimated 2 years
  correlation
Exploratory outcome:Clinical markers/ biomarkers as the potential predictive factor for regorafenib treatment outcome in overall cohort and long-term responders, assessed by changes in carbohydrate antigen (CA19-9) levels | through study completion, estimated 2 years
  correlation
Exploratory outcome: Image pattern as the potential predictive factor for regorafenib treatment outcome in overall cohort and long-term responders, assessed by changes in image patterns | through study completion, estimated 2 years
  correlation

CONTACTS AND LOCATIONS:
Overall Officials: Hao-Wei Teng, MD, PhD, Principal Investigator — Taipei Veterans General Hospital, Taiwan
Locations (1):
- Taipei Veterans General Hospital, Taipei, Taiwan

REFERENCES:
- [Derived] Hsu HC, Huang KC, Chen WS, Jiang JK, Yang SH, Wang HS, Chang SC, Lan YT, Lin CC, Lin HH, Huang SC, Cheng HH, Yang TS, Chen CC, Chao Y, Teng HW. Preference criteria for regorafenib in treating refractory metastatic colorectal cancer are the small tumor burden, slow growth and poor/scanty spread. Sci Rep. 2021 Jul 28;11(1):15370. doi: 10.1038/s41598-021-94968-x. PMID 34321583